CLINICAL TRIAL: NCT00918346
Title: Pharmacodynamics of Tafluprost 0.0015% Eye Drops: a Comparison Between the Preserved and Unpreserved Formulation in Patients With Open-angle Glaucoma or Ocular Hypertension
Brief Title: Pharmacodynamics of Tafluprost 0.0015% Eye Drops: a Comparison Between the Preserved and Unpreserved Formulation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santen Oy (Industry)
Responsible Party: Auli Ropo, MD, PhD, Santen Oy
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 77550
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Results first posted 2009-09-15 (Estimated); Last update posted 2010-12-28 (Estimated); Status verified 2010-12

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: Ocular hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tafluprost 0.0015% preserved formulation (Experimental)
  Interventions: Drug: Tafluprost 0.0015%
- Tafluprost 0.0015% unpreserved formulation (Experimental)
  Interventions: Drug: Tafluprost 0.0015%

INTERVENTIONS:
Drug: Tafluprost 0.0015% — Eye drops, 0.015 mg/ml, once daily to affected eye(s)

SUMMARY:
The objective of this study is to investigate the pharmacodynamics (as expressed in intraocular pressure [IOP]) of two formulations of tafluprost 0.0015% eyedrops (preserved and unpreserved) in patients with open-angle glaucoma or ocular hypertension.

The primary aim of this study is to show that IOP reduction between the two formulations is equivalent at the end of the 4 week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or more
* A diagnosis of open angle glaucoma or ocular hypertension
* Prior use of prostaglandin(s)
* Intra ocular pressure of 22-34 mmHg in at least one eye

Exclusion Criteria:

* Females who are pregnant, nursing or planning a pregnancy, or females of childbearing potential who are not using a reliable method of contraception
* Previous participation in any clinical trial in which tafluprost was an investigational drug or use of contact lenses at screening or during the study
* Presence of any abnormality or significant illness that could be expected to interfere with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2005-09; Primary Completion 2006-03 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juhani Airaksinen, Prof., Principal Investigator — University Hospital of Oulu
Locations (3):
- Oulu University Hospital, Oulu, Finland
- Germany (2):
  - Ulrich Richter's surgery, Regensburg
  - Praxis Dr. Hamacher, Starnberg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At 2 centers in Germany, 1 center in Finland:
  14 September 2005 first patient screened 08 November 2005 first patient randomized 05 April 2006 last patient completed
Pre-assignment Details: A total of 45 patients screened and 43 patients randomized. 2 screening failure patients: 1 withdrawn consent and 1 too low IOP (inclusion criterion 4).
Groups:
- Preserved Formulation First, Then Unpreserved Formulation: Tafluprost 0.0015% preserved formulation once daily for first 4 weeks, then unpreserved formulation (after washout)
- Unpreserved Formulation First, Then Preserved Formulation: Tafluprost 0.0015% unpreserved formulation once daily for first 4 weeks, then preserved formulation (after washout)
Period: First Treatment Period (4 Weeks)
Arm/Group | Preserved Formulation First, Then Unpreserved Formulation | Unpreserved Formulation First, Then Preserved Formulation
Started | 21 | 22
Completed | 21 | 21 (A patient completed the first treatment period but discontinued thereafter (did not start washout).)
Not Completed | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Period: Washout (at Least 4 Weeks)
Arm/Group | Preserved Formulation First, Then Unpreserved Formulation | Unpreserved Formulation First, Then Preserved Formulation
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0
Period: Second Treatment Period (4 Weeks)
Arm/Group | Preserved Formulation First, Then Unpreserved Formulation | Unpreserved Formulation First, Then Preserved Formulation
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0
Period: Post Study Period
Arm/Group | Preserved Formulation First, Then Unpreserved Formulation | Unpreserved Formulation First, Then Preserved Formulation
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes all 43 randomized patients (86 eyes)
Arm/Group | Entire Study Population
Number analyzed (Participants) | 43
Age Continuous [Mean (Standard Deviation); unit: years] | 65.3 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 16
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 43
Region of Enrollment [Number; unit: participants]
  Germany | 32
  Finland | 11
Diagnosis - worse eyes [Number; unit: eyes] — Worse eye: If both eyes satisfied the inclusion criteria, then the worse eye was the eye with the higher intraocular pressure at the 8:00 IOP measurement at the first baseline visit. In case both eyes had the same IOP, then the right eye was designated as the worse eye. If only one eye satisfied the inclusion criteria, then that eye was considered to be the worse eye.
  eyes
    Primary Open Angle Glaucoma | 28
    Capsular Glaucoma | 3
    Ocular Hypertension | 12
Central corneal thickness [Mean (Standard Deviation); unit: micrometer]
  Right eye | 548.7 (42.8)
  Left eye | 547.0 (45.4)

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressures (IOPs) at Baseline
Description: IOPs at baseline: mean IOP values at four timepoints (worse eye)
Time Frame: Baseline
Population: IOPs of all subjects who received preserved/unpreserved formulation
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Preserved Formulation: tafluprost 0.0015% preserved formulation
- Unpreserved Formulation: tafluprost 0.0015% unpreserved formulation
Arm/Group | Preserved Formulation | Unpreserved Formulation
Number analyzed (Participants) | 42 | 43
mmHg
  8 o'clock | 22.57 (3.04) | 22.98 (3.18)
  12 o'clock | 20.86 (2.79) | 21.78 (2.68)
  16 o'clock | 21.73 (3.19) | 21.51 (2.49)
  20 o'clock | 21.77 (3.02) | 21.81 (2.61)

2. Secondary Outcome: Overall and Time-wise Comparisons of IOP at Week 1
Description: The overall and time-wise, i.e. at 8:00, 12:00, 16:00 and 20:00, comparisons of IOP at week 1 (diurnal IOP and IOP value at given timepoint at 1 week minus corresponding value at baseline: unpreserved-preserved) were done using the RM ANCOVA model.
Time Frame: Baseline - Week 1
Population: ITT: randomized patients who received at least one dose of study medication and had at least one pharmacodynamic (IOP) measurement available.
Measure: Mean (95% Confidence Interval); unit: mmHg
Groups:
- RM ANCOVA: ITT Efficacy Dataset: randomized and received study medication
Arm/Group | RM ANCOVA: ITT Efficacy Dataset
Number analyzed (Participants) | 43
mmHg
  Overall | -0.27 [-0.73 to 0.19]
  Timepoint 8:00 | -0.32 [-0.96 to 0.32]
  Timepoint 12:00 | -0.25 [-0.89 to 0.40]
  Timepoint 16:00 | -0.39 [-1.03 to 0.26]
  Timepoint 20:00 | -0.13 [-0.77 to 0.52]

3. Secondary Outcome: Change From Baseline in Time-wise IOPs at Week 4
Description: The time-wise, i.e. at 8:00, 12:00, 16:00 and 20:00, comparisons of IOP at week 4 (IOP value at given timepoint at 4 weeks minus corresponding value at baseline: unpreserved-preserved) were done using the RM ANCOVA model.
Time Frame: Baseline - Week 4
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | RM ANCOVA: ITT Efficacy Dataset
Number analyzed (Participants) | 43
mmHg
  Timepoint 8:00 | 0.24 [-0.51 to 0.98]
  Timepoint 12:00 | 0.11 [-0.64 to 0.86]
  Timepoint 16:00 | 0.00 [-0.74 to 0.75]
  Timepoint 20:00 | -0.30 [-1.04 to 0.45]

4. Primary Outcome: Intraocular Pressures (IOPs) at Week 1
Description: IOPs at week 1: mean IOP values at four timepoints (worse eye)
Time Frame: Week 1
Population: IOPs of all subjects who received preserved/unpreserved formulation
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Preserved Formulation | Unpreserved Formulation
Number analyzed (Participants) | 42 | 43
mmHg
  8 o'clock | 16.43 (2.11) | 16.21 (2.70)
  12 o'clock | 15.77 (1.60) | 15.72 (1.92)
  16 o'clock | 16.23 (1.73) | 15.83 (1.99)
  20 o'clock | 16.26 (2.20) | 16.16 (2.08)

5. Primary Outcome: Intraocular Pressures (IOPs) at Week 4
Description: IOPs at week 4: mean IOP values at four timepoints (worse eye)
Time Frame: Week 4
Population: IOPs of all subjects who received preserved/unpreserved formulation
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Preserved Formulation | Unpreserved Formulation
Number analyzed (Participants) | 42 | 43
mmHg
  8 o'clock | 16.39 (2.43) | 16.80 (3.00)
  12 o'clock | 16.30 (2.46) | 16.67 (2.54)
  16 o'clock | 16.64 (2.37) | 16.71 (2.53)
  20 o'clock | 17.21 (1.91) | 17.01 (2.44)

6. Primary Outcome: Primary Pharmacodynamic Variable Intention to Treat Efficacy Dataset: Change From Baseline in the Overall Diurnal Intraocular Pressure (IOP) at Week 4 (Worse Eye)
Description: Overall treatment difference at 4 weeks (unpreserved-preserved) evaluated using a repeated measurements analysis of covariance (RM ANCOVA) model.
Time Frame: Baseline - Week 4
Population: Intention To Treat (ITT): randomized patients who received at least one dose of study medication and had at least one pharmacodynamic (IOP) measurement available.
Measure: Mean (95% Confidence Interval); unit: mmHg
Groups:
- RM ANCOVA: ITT Efficacy Dataset: randomized who received at least one dose of study medication and had at least one IOP measurement
Arm/Group | RM ANCOVA: ITT Efficacy Dataset
Number analyzed (Participants) | 43
mmHg | 0.01 [-0.46 to 0.49]
Statistical Analysis 1: Comparison: RM ANCOVA: ITT Efficacy Dataset; H1 (the alternative hypothesis aimed to be proven): the unpreserved formulation is equivalent with the preserved formulation; Test type: Non-Inferiority or Equivalence — The equivalence limit was set to 1.5 mmHg. Equivalence was shown if the two-sided 95% confidence interval for the difference (unpreserved-preserved) lay entirely within the equivalence range (-1.5 mmHg, 1.5 mmHg). Target sample size was 34 evaluable patients (40 randomized), assuming a standard deviation of 3.0 mmHg change in IOP, a power of 80%, an intra-class correlation coefficient of 0.60 and a twosided type 1 error rate of 5%; p = 0.96, ANCOVA; Baseline IOP a covariate; Mean Difference (Final Values) = 0.01, 95% CI [-0.46 to 0.49] — Analysis model used IOP measurements at four timepoints (at 8, 12, 16 and 20 o'clock) on Baseline and Week 4

7. Primary Outcome: Primary Pharmacodynamic Variable Per Protocol Efficacy Dataset: Change From Baseline in the Overall Diurnal Intraocular Pressure (IOP) at Week 4 (Worse Eye)
Description: Overall treatment difference at 4 weeks (unpreserved-preserved) evaluated using a repeated measurments analysis of covariance (RM ANCOVA) model.
Time Frame: Baseline - Week 4
Population: Per Protocol (PP): randomized patients who completed the study per protocol (i.e. excluded from PP is the discontinued patient and a patient with major protocol violation)
Measure: Mean (95% Confidence Interval); unit: mmHg
Groups:
- RM ANCOVA: PP Efficacy Dataset: randomized patients who completed the study per protocol (PP)
Arm/Group | RM ANCOVA: PP Efficacy Dataset
Number analyzed (Participants) | 41
mmHg | -0.05 [-0.52 to 0.42]
Statistical Analysis 1: Comparison: RM ANCOVA: PP Efficacy Dataset; [analysis description as in outcome 6, analysis 1]; Test type: Non-Inferiority or Equivalence — The equivalence limit was set to 1.5 mmHg. Equivalence was shown if the two-sided 95% confidence interval for the difference (unpreserved-preserved) lay entirely within the equivalence range (-1.5 mmHg, 1.5 mmHg). Target sample size was 34 evaluable patients (40 randomized), assuming a standard deviation of 3.0 mmHg change in IOP, a power of 80%, an intra-class correlation coefficient of 0.60 and a twosided type I error rate of 5%; p = 0.83, ANCOVA; Baseline IOP a covariate; Median Difference (Final Values) = -0.05, 95% CI [-0.52 to 0.42] — Analysis model used IOP measurements at four timepoints (at 8, 12, 16 and 20 o'clock) on Baseline and Week 4

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at Week 1 and Week 4 visits of treatment period I and II, as well as on last Post-study visit. Additionally, baseline symptoms were queried on Day 0 (=Baseline) visit of the two treatment periods.
Description: Patients were asked about ocular or non-ocular symptoms with a non-leading question, or they volunteered the information during a study visit. Also, any clinically significant signs observed by the investigator could be recorded as adverse events.
Groups:
- Preserved Formulation: Tafluprost 0.0015% preserved formulation once daily for 4 weeks
- Unpreserved Formulation: Tafluprost 0.0015% unpreserved formulation once daily for first 4 weeks
Arm/Group | Preserved Formulation | Unpreserved Formulation
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/43
Other Adverse Events (participants affected / at risk) | 7/42 | 11/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preserved Formulation (N=42) | Unpreserved Formulation (N=43)
Conjunctival hyperemia (Eye disorders) | 2 (2) | 6 (6)
Ocular hyperemia (Eye disorders) | 0 (0) | 2 (2)
Erythema of eyelid (Eye disorders) | 1 (1) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1) | 1 (1)
Foreign body sensation (Eye disorders) | 1 (1) | 1 (1)
Anterior chamber cell (Eye disorders) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1)
Punctate keratitis (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Asthenopia (Eye disorders) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Superficial injury of eye (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor respects the investigators' wish to publish results of the study, and will not unnecessarily restrict the spreading of information of scientific interest. However, the study may involve confidential information affecting the company's business, such as aspects related to patent application. Therefore, the investigators agree to allow the sponsor to review any manuscripts and to negotiate timing and forum of publication.